CLINICAL TRIAL: NCT04467398
Title: Incidence of Intravascular (IV) Injection During Trigeminal Nerve Blocks and Impact of Needle Types to the IV Uptake: A Prospective Cohort Study
Brief Title: Incidence of Intravascular (IV) Injection During Trigeminal Nerve Blocks
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University (Other)
Responsible Party: Principal Investigator, Jeeyoun Moon, Associate Professor, Seoul National University
Other Study IDs: 2004-207-1120
Record Dates: First submitted 2020-05-22; First posted 2020-07-13 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Trigeminal Neuralgia; Facial Pain; Postherpetic Neuralgia; Cluster Headache
MeSH Terms: conditions — Trigeminal Neuralgia; Facial Pain; Neuralgia, Postherpetic; Cluster Headache

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tuohy needle group: The participants who undergo the trigeminal nerve block using 22 guage Tuohy needle.
  Interventions: Procedure: trigeminal nerve block
- Quincke needle group: The participants who undergo the trigeminal nerve block using 22 guage Quincke needle.
  Interventions: Procedure: trigeminal nerve block

INTERVENTIONS:
Procedure: trigeminal nerve block — Trigeminal nerve or branch block using 22 gauge Quincke or Tuohy needle under fluoroscopic guidance.

SUMMARY:
The purpose of this study is to investigate the incidence of intravascular injection during trigeminal nerve blocks.

DETAILED DESCRIPTION:
The patients who already scheduled for trigeminal nerve blocks will be randomized in a 1:1 ratio to tuohy needle group or quincke needle group after being informed about the study.

ELIGIBILITY:
Inclusion Criteria:

* The patients who scheduled to undergo trigeminal nerve block due to the facial pain

Exclusion Criteria:

* Refusal of the patient
* Pregnancy
* Coagulopathy
* Local or systemic infection
* Allergy to injectate
* Anatomical deformation of the skull

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who scheduled to undergo trigeminal nerve block because of:
  1. Trigeminal neuralgia/neuropathy
  2. Postherpetic trigeminal neuralgia
  3. Atypical facial pain
  4. Cluster headache
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-07-20 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
IV uptake prevalence (%) | During the procedure
  The incidence of intravascular injection during the procedure by digital subtraction angiography(DSA).

SECONDARY OUTCOMES:
Difference in incidence of intravascular injection | During the procedure
  Difference in incidence of intravascular injection according to needle type by DSA.
Total incidence of blood aspiration | During the procedure
  Total incidence of blood aspiration by regurgitation.
Total incidence of intravascular injection | During the procedure
  Total incidence of intravascular injection under non-DSA technique.
The depth of inserted needle when the practitioner check the intravascular uptake under DSA technique. | During the procedure
  The depth of inserted needle when the practitioner check the intravascular uptake under SDA technique.
The number of needle adjustment. | During the procedure
  The number of needle adjustment due to the intravascular uptake.
Total volume of local anesthetics for skin anesthesia. | During the procedure
  Total volume of local anesthetics for skin anesthesia.
Time for the procedure. | During the procedure
  Time for the procedure.
Total amount of radiation exposure for the procedure. | During the procedure
  Total amount of radiation exposure for the procedure.
Laterality | During the procedure
  The difference in incidence by the lateriality.
Final pattern of the fluoroscopic image | During the procedure
  The quality of the image(3: excellent, 2: acceptable, 1: not relevant)
Post-procedure pain | Within 1 hour after the procedure.
  NRS pain score after the procedure in recovery room
The difficulty of the procedure | Within 1 hour after the procedure.
  The difficulty grade by the practitioner(5:very easy, 4: relatively easy, 3:so so, 4:somewhat difficult, 1:very difficult)
The difference in incidence of blood aspiration | During the procedure.
  Difference in incidence of intravascular injection according to needle type by regurgitation.
The difference in incidence of intravascular injection. | During the procedure
  Difference in incidence of intravascular injection according to needle type by non-DSA technique.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No